CLINICAL TRIAL: NCT05528419
Title: Sacubitril Valsartan in Preventing the Recurrence of Atrial Fibrillation After Ablation in Elderly Hypertensive Patients With Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUPERIOR
Record Dates: First submitted 2022-09-02; First posted 2022-09-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation Recurrent; Hypertension
Keywords: elderly; ablation; blood pressure
MeSH Terms: conditions — Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Intervention Model Description: After screening period, eligible patients will be randomly assigned into sacubitril/valsartan group (sacubitril/valsartan 80mg QD) or valsartan group (valsartan 80mg QD).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril valsartan (Experimental)
  Interventions: Drug: Sacubitril-valsartan
- Valsartan (Active Comparator)
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Sacubitril-valsartan — sacubitril valsartan 100mg initiated, and titrated to 200mg according to mean clinic blood pressure at 1-month follow-up
  Arms: Sacubitril valsartan
Drug: Valsartan — valsartan 80mg initiated, and titrated to 160mg according to mean clinic blood pressure at 1-month follow-up
  Arms: Valsartan

SUMMARY:
Study name: Sacubitril Valsartan in Preventing the Recurrence of Atrial Fibrillation After Ablation in Elderly Hypertensive Patients With Atrial Fibrillation.

Medicine: sacubitril/valsartan (100mg) and valsartan (80mg).

Rationale: The latest guidelines represent an intensified management approach to reduce or prevent morbidity associated with atrial fibrillation. They provide stronger and more specific recommendations for catheter ablation (CA) use. However, not all patients maintain sinus rhythm after CA and both early and late relapses of AF can occur in many patients.

Objective: To evaluate the efficacy and safety of sacubitril/valsartan in preventing atrial fibrillation recurrences after ablation in elderly hypertensive patients with atrial fibrillation.

Study design: This is a 12-month prospective, randomized, active-controlled, open-label, multi-center study, with two treatment groups: sacubitril/valsartan (100mg tablet) and valsartan (80mg tablet).

Study population: Men or women aged between 55 and 80 years will be screened for hypertension. Eligible patients should be untreated and treated atrial fibrillation patients with clinic systolic/diastolic blood pressure ≥130/80 mmHg, who are going to receive catheter ablation procedure. Patients should have abilities to understand the study requirements and provide informed consent.

Randomization and treatment: After screening period by centers, eligible patients will be randomly divided into 2 groups, taking one pill of sacubitril/valsartan (100mg tablet) or valsartan (80mg tablet).

Follow-up: After meeting the inclusion criteria, there will be 1-week screening period. Clinic blood pressure, ambulatory blood pressure, echocardiography, concomitant medication records and adverse event records will be collected at randomization period. Then patients will be randomly assigned into sacubitril/valsartan group and valsartan group. The treatment will be observed for 12 months. There will be 4 visiting points in the treatment period, which will be the 1st month, 3rd month, 6th month and 12th month.

Sample size: A total of 320 patients should be enrolled in total.

Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital, recruitment will start. Patients enrollment and follow-up are expected to be performed from October 2022 to June 2026.

DETAILED DESCRIPTION:
Study name: Sacubitril Valsartan in Preventing the Recurrence of Atrial Fibrillation After Ablation in Elderly Hypertensive Patients With Atrial Fibrillation.

Medicine: sacubitril/valsartan (100mg) and valsartan (80mg).

Rationale: The latest guidelines represent an intensified management approach to reduce or prevent morbidity associated with atrial fibrillation. They provide stronger and more specific recommendations for catheter ablation (CA) use. However, not all patients maintain sinus rhythm after CA and both early and late relapses of AF can occur in many patients.

Objective: To evaluate the efficacy and safety of sacubitril/valsartan in preventing atrial fibrillation recurrences after ablation in elderly hypertensive patients with atrial fibrillation.

Study design: This is a 12-month prospective, randomized, active-controlled, open-label, multi-center study, with two treatment groups: sacubitril/valsartan (100mg tablet) and valsartan (80mg tablet).

Study population: Men or women aged between 55 and 80 years will be screened for hypertension. Eligible patients should be untreated and treated atrial fibrillation patients with clinic systolic/diastolic blood pressure ≥130/80 mmHg, who are going to receive catheter ablation procedure. Patients should have abilities to understand the study requirements and provide informed consent.

Randomization and treatment: After screening period by centers, eligible patients will be randomly divided into 2 groups, taking one pill of sacubitril/valsartan (100mg tablet) or valsartan (80mg tablet).

Follow up: After meeting the inclusion criteria, there will be 1-week screening period. Clinic blood pressure, ambulatory blood pressure, echocardiography, concomitant medication records and adverse event records will be collected at randomization period. Then patients will be randomly assigned into sacubitril/valsartan group and valsartan group. The treatment will be observed for 12 months. There will be 4 visiting points in the treatment period, which will be the 1st month, 3rd month, 6th month and 12th month.

Sample size: A total of 320 patients should be enrolled in total.

Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital, recruitment will start. Patients enrollment and follow-up are expected to be performed from October 2022 to June 2026.

Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 55-80;
2. Persistent ot paroxysmal atrial fibrillation patients who are going to receive catheter ablation surgery;
3. Clinic systolic blood pressure (SBP) ≥ 130 or diastolic blood pressure (DBP) ≥ 80 mmHg) in untreated and treated patients；
4. Ability to understand the study requirements and provide informed consent.

Exclusion Criteria:

1. Secondary hypertension;
2. Clinic SBP/DBP≥180/110 mmHg, or 24-h ambulatory mean SBP/DBP<120/70 mmHg;
3. Coronary heart disease, valvular heart disease, hypertrophic cardiomyopathy, pulmonary heart disease, hyperthyroidism or hypothyroidism;
4. New York Heart Association functional class IV, or left ventricular ejection fraction of <30%;
5. Implanted pacemaker or defibrillator, myocardial infarction or percutaneous coronary intervention of ≤ 6 months before ablation;
6. Presence of LA thrombus on transesophageal echocardiography;
7. Severe hepatic or severe renal dysfunction estimated glomerular filtration rate of < 30 mL/min*per1.73 m2;
8. Serum potassium >5.5 mmol/L;
9. Pregnant or lactating women;
10. Other circumstances that patients are not appropriate for the study upon the investigator's judgment;
11. Patients who are receiving other study drugs or study medical devices;
12. Unwilling or unable to provide informed consent.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
Any documented atrial arrhythmia (AF, atrial flutter, or atrial tachycardia) episode lasting for at least 30 s after a 3-month blanking period | 3-12 months

SECONDARY OUTCOMES:
Any documented atrial arrhythmia (AF, atrial flutter, or atrial tachycardia) episode lasting for at least 30 s within the 3-month blanking period. | 0-3 months
Change in mean office and ambulatory blood pressure after 12-month treatment from baseline in each group | Baseline and 12 months
Change in NT-proBNP after 12-month treatment from baseline in each group | Baseline and 12 months
Change in left atrial GLS from echocardiograph after 12-month treatment from baseline in each group | Baseline and 12 months
Change in mean office blood pressure after 3-month treatment from baseline in each group | Baseline and 3 months
Change in NT-proBNP after 3-month treatment from baseline in each group | Baseline and 3 months
Change in left atrial GLS from echocardiograph after 3-month treatment from baseline in each group | Baseline and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China